CLINICAL TRIAL: NCT00593216
Title: New Diagnosis Of Vestibular Vertigo With Functional MRI
Brief Title: Diagnosis Of Vertigo With New Imaging
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Kenneth Grundfast M.D., Department of Surgery-Otolaryngology of Boston University Medical Center
Other Study IDs: H-25852
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Vertigo
Keywords: functional magnetic Resonance Imaging; vertigo; vestibular
MeSH Terms: conditions — Vertigo | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Healthy volunteers devoid of any ear problems
  Interventions: Device: Functional MRI imaging
- Vertigo: Patients with the symptoms of vertigo
  Interventions: Device: Functional MRI imaging

INTERVENTIONS:
Device: Functional MRI imaging — The functional MRI imaging of whole brain will be obtained before, during and after the vestibular response which is induced by the designated caloric stimulation. Post-imaging analysis will reveal which region or neural pathways in the central nervous system may attributed to the development of vertigo.
  Other Names: Magnetic Resonance Imaging

SUMMARY:
The purpose of this study is to determine the potential usefulness of new functional MRI in diagnostic assessment of patients presenting with vertigo.

DETAILED DESCRIPTION:
The incidence of vertigo has been reported to be as high as 1.5% in the general population and some reports suggest that more than 5% of adults experience some kind of vertigo each year. In 80% of affected individuals, this symptom resulted in a medical consultation, interruption of daily activities, or sick leave. Therefore, vertigo can have a significant impact on health and well being. Unfortunately, there is not yet any satisfactory objective method for diagnosis of vertigo. At present, the diagnosis usually depends on medical history, vestibular function tests, Dix-Hallpike positioning tests done in the office, and, to some extent imaging studies doen to look for such abnormalities such as acoustic tumor, brain tumor, and evidence of multiple sclerosis. A number of recent studies support the possibility of using functional MRI (fMRI), particularly a new diffusion tensor fiber tracking (DTT) technique, as a new tool for diagnosis of disorders that can cause vertigo. In this study, our hypothesis is that there is an alteration in the activity in neural pathways of patients with vertigo that can be detected by fMRI. To test this assumption, our objective in this study is to determine whether there is a difference between the fMRI images obtained in normal subjects versus those in patients with vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer or patient with symptom of vertigo

Exclusion Criteria:

* Evidence of mental impairment
* Any type of bioimplant or any type of ferromagnetic bioimplant
* Pregnant females
* Exhibit noticeable anxiety and/or claustrophobia
* History of serious disease in central nervous and cerebrovascular systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Activation of target sites on the functional MRI images during the vestibular response | Not specific

SECONDARY OUTCOMES:
Differences in the fiber tracking of central nervous system specifically involved in the vestibular response | Not specific

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Grundfast, M.D., Principal Investigator — Department of Otolaryngology- Head and Neck surgery of Boston University Medical Center